CLINICAL TRIAL: NCT06614959
Title: Assessing the Effects of Oscillatory Positive Expiratory Pressure (OPEP) Therapy on Disease Impact and Respiratory System Dynamics in Patients With COPD: A Prospective Non-Pharmacologic Interventional Cohort Study
Brief Title: The Effects of Oscillatory Positive Expiratory Pressure (OPEP) Therapy in Patients With COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Trudell Medical International (Industry)
Responsible Party: Principal Investigator, Bryan A. Ross, Clinician-Scientist (RI-MUHC), Respirologist (MUHC), Assistant Professor (McGill University), McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-10838
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: COPD
Keywords: COPD; OPEP; Chronic Bronchitis; Disease Impact; Reactance; CASA-Q Questionnaire; Oscillometry
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oscillatory Positive Expiratory Pressure (OPEP) therapy arm (Experimental): Participants will receive and use the smart OPEP device at least twice a day in the home environment for 4 consecutive weeks.
  Interventions: Device: Oscillatory Positive Expiratory Pressure (OPEP) Therapy

INTERVENTIONS:
Device: Oscillatory Positive Expiratory Pressure (OPEP) Therapy — The smart OPEP device is a standard OPEP device equipped with an additional detachable sensor that collects diagnostic information on the total elapsed time of OPEP use, the pressure generated during use, frequency and amplitude of pressure oscillations, respiratory information (inhalations/exhalation number/time), and sum of all oscillations with a pressure over 1 centimeter of water (cmH2O), all of which will inform the duration and quality of home use.

SUMMARY:
The goal of this non-pharmacologic interventional study is to learn if Oscillatory Positive Expiratory Pressure (OPEP) therapy can improve disease impact and respiratory system dynamics in patients with COPD. The main questions it aims to answer are:

Is OPEP therapy able to improve the impact of cough symptoms as measured on a validated symptom score? Is OPEP therapy able to improve the properties of the lung (called reactance) as measured by oscillometry?

Researchers will compare the results of the same tests performed before and after 4 weeks of OPEP treatment to see if OPEP treatment improves cough symptoms and lung mechanics.

* Participants with COPD will complete in-person baseline tests and will then receive the smart OPEP device.
* These participants will then use the smart OPEP device at home, at least twice a day, for 4 consecutive weeks.
* Finally, these participants will return to complete in-person end-of-study tests.

DETAILED DESCRIPTION:
The objectives of this prospective, non-pharmacologic interventional cohort study are to determine the effect of four consecutive weeks of twice-daily or greater OPEP usage among patients with COPD with a chronic bronchitis (sputum-producing) phenotype on disease impact and on respiratory system dynamics. A 'dose-response' effect of OPEP use will also be investigated.

We hypothesize that a 4-week period of OPEP therapy among eligible patients with COPD with a chronic bronchitis (sputum-producing) phenotype will be associated with improved disease impact scores and airway mechanics.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 40 years of age or more
2. Former/current smokers with a cigarette smoking history for 10 or more pack-years
3. Physician diagnosis of COPD previously confirmed by spirometry (FEV1/FVC less than 0.7) with 'mild' to 'very severe' (i.e. GOLD 1-4) COPD
4. Chronic bronchitis phenotype: Sputum production or presence of productive cough greater than 2 days/week in the last 3 months for at least 2 consecutive years, or presence of cough and phlegm almost every day or several times per week
5. Ability to participate without supplemental oxygen during all oscillometry testing
6. Ability to provide informed consent

Exclusion Criteria:

1. No COPD diagnosis
2. Bronchiectasis, cystic fibrosis, or any other known suppurative acute/chronic lung disease as the principal respiratory condition
3. Physician-diagnosed exacerbation and/or hospitalization for pulmonary symptoms in the 4 weeks preceding baseline testing
4. Current use of OPEP, or any use of OPEP in the 4 weeks preceding baseline testing
5. Current or recent participation in a standard Pulmonary Rehabilitation program in the 4 weeks preceding baseline testing or during the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Cough Impact Domain of the CASA-Q (co-primary outcome) | Baseline (within 7 days preceding the 4-week intervention period) and End-of-Study (within 7 days following the 4-week intervention period).
  The Cough and Sputum Assessment Questionnaire (CASA-Q) is a validated tool used to assess cough and sputum symptoms in patients with COPD and has been shown to be responsive to changes in these aspects during clinical trials, and following exacerbations. 20-item questionnaire consisting of four domains. The magnitude of difference in baseline and end-of-study visit 'Cough Impact' domain from the CASA-Q score will serve as the co-primary outcome for disease impact.
Reactance at 5 Hertz (Hz) (co-primary outcome) | Baseline (within 7 days preceding the 4-week intervention period) and End-of-Study (within 7 days following the 4-week intervention period).
  Oscillometry can detect changes in respiratory system resistance and reactance as well as flow-limited breaths. The magnitude of difference in baseline and end-of-study visit reactance of the respiratory system at 5 Hz (X5) will serve as the co-primary outcome for respiratory system dynamics.

SECONDARY OUTCOMES:
COPD Assessment Test (CAT) | Baseline (within 7 days preceding the 4-week intervention period) and End-of-Study (within 7 days following the 4-week intervention period).
  The CAT is a validated self-administered questionnaire that is used for assessing and monitoring symptom burden and health-related quality of life in patients with COPD.
Sputum Impact | Baseline (within 7 days preceding the 4-week intervention period) and End-of-Study (within 7 days following the 4-week intervention period).
  Sputum Impact domain (6 items) of the CASA-Q Questionnaire.
The reactance-volume loop area (AXV) | Baseline (within 7 days preceding the 4-week intervention period) and End-of-Study (within 7 days following the 4-week intervention period).
  Measurement obtained from intra-breath oscillometry.
Mean inspiratory minus expiratory total respiratory system reactance (mean ∆Xrs) | Baseline (within 7 days preceding the 4-week intervention period) and End-of-Study (within 7 days following the 4-week intervention period).
  Measurement obtained from intra-breath oscillometry.
Area of reactance (Ax) | Baseline (within 7 days preceding the 4-week intervention period) and End-of-Study (within 7 days following the 4-week intervention period).
  Measurement obtained from oscillometry.
Resonant frequency (Fres) | Baseline (within 7 days preceding the 4-week intervention period) and End-of-Study (within 7 days following the 4-week intervention period).
  Measurement obtained from oscillometry.
Sputum Symptom Severity | Baseline (within 7 days preceding the 4-week intervention period) and End-of-Study (within 7 days following the 4-week intervention period).
  Sputum Symptom Severity Domain (3 items) of the CASA-Q Questionnaire
  .
Cough Symptom Severity | Baseline (within 7 days preceding the 4-week intervention period) and End-of-Study (within 7 days following the 4-week intervention period).
  Cough Symptom Severity Domain (3 items) of the CASA-Q Questionnaire.
Cough Impact | Baseline (within 7 days preceding the 4-week intervention period) and End-of-Study (within 7 days following the 4-week intervention period).
  Cough Impact Domain (8 items) of the CASA-Q Questionnaire.
The difference between resistance at 5 Hertz (R5) and resistance at 20 Hertz (R20) (R5-20) | Baseline (within 7 days preceding the 4-week intervention period) and End-of-Study (within 7 days following the 4-week intervention period).
  Measurement obtained from oscillometry.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan A. Ross, MD, MSc (Physiol), MSc (Epi), Principal Investigator — RI-MUHC/MUHC
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Due to data privacy regulations, individual participant data collected during this study is not publicly accessible. However, access to anonymized data may be granted upon evaluation. Additional documents will also be available upon inquiry. All requests should be directed to the corresponding author (BAR).